CLINICAL TRIAL: NCT06877026
Title: Evaluating the Repeatability and Reproducibility of FibroScan Generations
Brief Title: FibroScan-Reproducibility and Repeatability Study
Acronym: FibroScan-RR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Echosens (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: M141
Record Dates: First submitted 2025-01-17; First posted 2025-03-14 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Liver Disease; Alcohol-Related
Keywords: FibroScan; Reproducibility; Repeatability
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Full Cohort (Experimental): This population will be defined by patients fulfilling all inclusion and exclusion criteria.
  Interventions: Device: FibroScan; Other: Liver Enzymes

INTERVENTIONS:
Device: FibroScan — Day 1 = 5 FibroScan examinations Day 2 = 4 FibroScan examinations
Other: Liver Enzymes — Day = 1 blood collection for liver enzymes. Day 2= 1 blood collection for liver enzymes.

SUMMARY:
Chronic liver disease (CLD) is a serious health issue worldwide, often progressing without symptoms until advanced stages with risks of complications like liver cancer and cirrhosis. Early detection is crucial to help prevent these outcomes. Liver stiffness measurement (LSM) can detect fibrosis (scarring) in the liver, a common issue in CLD patients while traditional methods like liver biopsy are invasive and not ideal for regular screening and monitoring.

FibroScan, a non-invasive device, measures the liver stiffness and fat content in the liver. This study will assess how reliable and consistent FibroScan results are when used by different operators and across different days, focusing on patients with liver conditions like metabolic-related liver disease (MASLD), alcohol-related liver disease (ALD), and hepatitis B. This research also aims to test both the standard and Guided VCTE (Vibration Controlled Transient Elastography) FibroScan generations to evaluate their reproducibility and repeatability. As secondary objectives the Control Attenuation Parameter (CAP) results, and the FAST, Agile 3+, and Agile 4 scores will be evaluated to compare their reproducibility and repeatability.

Adult participants will attend two visits within three days. During these visits, they will undergo multiple FibroScan scans that include five scans on Day 1 (visit 1) and four scans on the follow up visit (visit 2), one blood sample for liver health assessment on each visit, and an AUDIT questionnaire on Day 1 (visit 1). Some participants may undergo only two scans on the follow-up visit since this will depend on operator availability. Each session will last 25-45 minutes including all examination types.

The study is funded by Echosens, the manufacturer of FibroScan, and will be conducted at UK healthcare facilities in England. By evaluating the variability of FibroScan results, this research could lead to a better understanding of the device's reproducibility and reliability in measuring liver stiffness across different operators and time points, potentially enhancing clinical confidence in its use for managing chronic liver diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥ 18 y.o) with Metabolic Dysfunction Associated Steatotic Liver Disease (MASLD), Metabolic and Alcohol-related Liver Disease (MetALD), and Alcohol-related Liver Disease (ALD).
* Adult patients able to give written informed consent.

Exclusion Criteria:

* Vulnerable patients
* Patients with other chronic liver disease including but not limited to hepatitis B, hepatitis C, autoimmune hepatitis, cholestatic diseases
* Patients with ascites
* Patients with elevated conjugated bilirubin (>1.5 ULN)
* Patients with heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine if guided VCTE, as opposed to a standard examination, improves LSM reproducibility across different days and different operators. | From Day 1 (first visit) to Day X (follow up visit, Day X can be up to 3 days after Day 1visit).
  Reproducibility of LSM by Guided VCTE versus standard examination, when performed on different days and by different operators. Day 1 is the first visit and Day X is the follow up visit. Day X can be up to 3 days after the Day 1 visit.

SECONDARY OUTCOMES:
To determine if guided VCTE, as opposed to a standard examination, improves CAP, FAST, Agile 3+ and Agile 4 reproducibility across different days and different operators. | From Day 1 (first visit) to Day X (follow up visit, Day X can be up to 3 days after Day 1visit)
  Reproducibility of CAP, FAST, Agile 3+ and Agile 4 by Guided VCTE versus standard examination, when performed on different days (Day 1 and Day X, X≤ 3 calendar days after Day 1) and by different operators
To determine if guided VCTE, as opposed to a standard examination, improves LSM and CAP, FAST, Agile 3+ and Agile 4 reproducibility across different days with the same operator. | From Day 1 (first visit) to Day X (follow up visit, Day X can be up to 3 days after Day 1visit)
  Reproducibility of LSM and CAP, FAST, Agile 3+ and Agile 4 by Guided VCTE versus standard examination, when performed on different days (Day 1 and Day X, X≤ 3 calendar days after Day 1) by the same operator
To determine if guided VCTE, as opposed to a standard examination, improves LSM and CAP, FAST, Agile 3+ and Agile 4 repeatability on the same day with the same operator | Day 1 only (1st visit only)
  Repeatability of LSM and CAP, FAST, Agile 3+ and Agile 4 by Guided VCTE versus standard examination, when performed on the same day (Day 1 only) and by the same operator
To evaluate the effect of resting time vs no resting time before the FibroScan Standard examination for both LSM and CAP. | Day 1 only (1st visit only)
  Repeatability of LSM and CAP, FAST, Agile 3+ and Agile 4 by Guided VCTE with (5 minutes) or without resting time and with or without control breathing performed on the same day (Day 1 only) by the same operator

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No